CLINICAL TRIAL: NCT04132947
Title: MET-REPAIR CONVAL: Concurrent Validity of the MET-REPAIR Questionnaire in German and of the Duke Activity Scale Index for Estimating Exercise Capacity Measured Using Exercise Testing
Brief Title: Validity of the MET-REPAIR Questionnaire
Acronym: MET-REPAIR Val
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01930
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Cohort Study correlating self reported exercise activity and spiroergometry results

SUMMARY:
MET-REPAIR CONVAL is an international cohort study to examine the ability of self-reported exercise capacity to predict perioperative cardiovascular events correcting for preoperative risk factors.

ELIGIBILITY:
Inclusion Criteria:

* over 45 years of age
* clinically indicated exercise testing
* signed written informed consent

Exclusion Criteria:

* unable to complete the questionnaire
* unable to consent or unwilling to participate
* cancelled exercise

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admitted to the ambulatory cardiology ward
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Metabolic equivalents (METs) | at Baseline
  METs per spiroergometry; assessment at time of clinically mandated spiroergometry

CONTACTS AND LOCATIONS:
Overall Officials: Eckhard Mauermann, Dr. med. MD, Principal Investigator — University Hospital Basel, Dep. of Anesthesia
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No